CLINICAL TRIAL: NCT00604968
Title: Caelyx(R) in Breast Cancer in the Elderly. Pegylated Liposomal Doxorubicin (Caelyx(R)) as Monotherapy in Elderly Patients With Locally Advanced and/or Metastatic Breast Cancer.
Brief Title: Pegylated Liposomal Doxorubicin (Caelyx(R)) as Monotherapy in Elderly Patients With Locally Advanced and/or Metastatic Breast Cancer (Study P05059)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05059
Record Dates: First submitted 2008-01-21; First posted 2008-01-30 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caelyx (Experimental)
  Interventions: Drug: Caelyx (pegylated liposomal doxorubicin; SCH 200746)

INTERVENTIONS:
Drug: Caelyx (pegylated liposomal doxorubicin; SCH 200746) — Caelyx will be administered intravenously at a dose of 40 mg/m^2 on day one every 4 weeks until progression, or unacceptable toxicity, or other reason to discontinue the study treatment. The drug is diluted in 250 ml glucose 5% (500 ml for doses >=90 mg).

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of pegylated liposomal doxorubicin (Caelyx) in elderly patients who are to receive first-line chemotherapy for metastatic or locally advanced breast cancer, not amenable to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the following criteria will be eligible for enrollment.

  * Female patients with histologic or cytologic diagnosis of breast cancer that is locally advanced or metastatic, and not amenable to surgery.
  * Age >= 65 years.
  * World Health Organization (WHO) Performance Status 0 - 2
  * Measurable disease in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Patients with bone metastasis can also be included but will be evaluated according to WHO criteria. Patients with non-measurable disease can also be included.
  * Left ventricular ejection fraction (LVEF) >= 50% verified by ultrasound cardiography (UCG); no clinical signs of heart disease.
  * Normal organ function, except due to disease involvement, however maximum deviation:

    * S-creatinine <= 1.5 x upper normal limit;
    * Bilirubin <= 2 x upper normal limit;
    * Alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) <= 3 x upper normal limit. In case of liver metastases, ALAT and/or ASAT <= 5 x upper normal limit.
  * Adequate bone marrow function, ie:

    * Platelets >= 100 x 10^9/L;
    * Neutrophils >= 1.5 x 10^9/L;
    * White Blood Cell (WBC) >= 3.0 x 10^9/L;
    * Hemoglobin > 90 g/L.
  * Life expectancy >= 12 weeks.
  * Patients having received oral and written information and having provided written informed consent.

Exclusion Criteria:

* Patients will not be enrolled if any of the following conditions apply.

  * Previous chemotherapy for metastatic disease. (The patient may have received previous endocrine therapy or single-drug Herceptin. Intrapleural or intrapericardial Novantrone is allowed.)
  * Recurrence <= 12 months after adjuvant anthracycline-containing treatment and/or prior doxorubicin > 300 mg/m^2 or epirubicin > 540 mg/m^2.
  * Myocardial infarction within 6 months of planned inclusion.
  * Symptomatic brain metastases.
  * Human Epidermal growth factor Receptor 2 (HER-2) positivity eligible for treatment with trastuzumab, or estrogen receptor (ER) positivity eligible for hormonal therapy.
  * Allergy to anthracyclines.
  * Uncontrolled infection.
  * Other not radically treated malignancy.
  * Other disease or condition contraindicating treatment or not allowing follow-up.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02-07 (Actual); Primary Completion 2009-10-16 (Actual); Study Completion 2009-10-16 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Green H, Stal O, Bachmeier K, Backlund LM, Carlsson L, Hansen J, Lagerlund M, Norberg B, Franzen A, Aleskog A, Malmstrom A. Pegylated liposomal doxorubicin as first-line monotherapy in elderly women with locally advanced or metastatic breast cancer: novel treatment predictive factors identified. Cancer Lett. 2011 Dec 27;313(2):145-53. doi: 10.1016/j.canlet.2011.07.017. Epub 2011 Aug 31. PMID 22056077

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 patients were screened and 25 were enrolled. All 25 patients enrolled received >=1 cycle of treatment with Caelyx. Per protocol, treatment was to continue until progression, unacceptable toxicity, or other reason for discontinuation of treatment - all subjects eventually discontinued treatment but were considered to have completed the study.
Groups:
- Caelyx: Caelyx was administered intravenously at a dose of 40 mg/m^2 on day one every 4 weeks until progression, or unacceptable toxicity, or other reason to discontinue the study treatment. The drug was diluted in 250 ml glucose 5% (500 ml for doses >=90 mg).
Period: Overall Study
Arm/Group | Caelyx
Started | 25
Completed | 25 (Due to the nature of study, all subjects receiving drug were considered to have completed.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Caelyx
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure (Defined as Progression of Disease [According to the Response Evaluation Criteria in Solid Tumors (RECIST) or World Health Organization (WHO) Criteria] or Unacceptable Toxicity Leading to Discontinuation of Treatment or Death).
Description: Treatment failure was defined as progression of disease (according to the RECIST or WHO criteria) or unacceptable toxicity leading to discontinuation of treatment or death. Progressive Disease according to RECIST response criteria: >=20% increase in the sum of the Longest Diameter of target lesions or unequivocal progression of non-target lesions. Appearance of new lesions will also constitute progressive disease. Progressive Disease according to WHO response criteria: Increase in size of existing lesions or appearance of new lesions.
Time Frame: Time of treatment until progression of disease or unacceptable toxicity leading to discontinuation of treatment or death, assessed every 12th week until end of treatment (study planned to continue until all participants ended treatment).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Caelyx
Number analyzed (Participants) | 25
Months | 5.52 [3.67 to 8.52]

2. Secondary Outcome: Number of Patients With Stable Disease (SD) as Best Response
Description: Response was calculated according to RECIST criteria except for bone metastasis where WHO criteria was used. For patients with skeletal disease only, WHO criteria was used. For patients with measurable disease according to RECIST as well as bone metastasis, both RECIST & WHO were used.
  RECIST response criteria for SD required steady state of response of at least 9 weeks duration. There may be no appearance of new lesions.
  WHO response criteria for SD required no significant change for at least 8 weeks.
Time Frame: Time of treatment until treatment discontinuation, assessed every 12th week until end of treatment (study planned to continue until all participants ended treatment).
Population: 10 patients were followed by RECIST, 4 patients were followed by WHO Response criteria, and 8 patients by both RECIST and WHO Response criteria (n=22). 3 patients had non-measurable disease and could not be included in the analysis.
Measure: Number; unit: participants
Arm/Group | Caelyx
Number analyzed (Participants) | 22
participants
  Patients followed by RECIST only (n=10) | 5
  Patients followed by WHO only (n=4) | 4
  Patients followed by RECIST & WHO (n=8) | 4

3. Secondary Outcome: Number of Patients With Partial Response (PR) as Best Response
Description: Response was calculated according to RECIST criteria except for bone metastasis where WHO criteria was used. For patients with skeletal disease only, WHO criteria was used. For patients with measurable disease according to RECIST as well as bone metastasis, both RECIST & WHO were used.
  RECIST PR criteria required >=30% decrease in certain target lesions & no increase in size of non-target lesions or appearance of new lesions
  WHO PR criteria required partial decrease in size of lytic lesions, recalcification of lytic lesions, or decreased density of blastic lesions for >=4 wks
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Caelyx
Number analyzed (Participants) | 22
participants
  Patients followed by RECIST only (n=10) | 1
  Patients followed by WHO only (n=4) | 0
  Patients followed by RECIST & WHO (n=8) | 2

4. Secondary Outcome: Number of Patients With Progressive Disease (PD) as Best Response
Description: Response was calculated according to RECIST criteria except for bone metastasis where WHO criteria was used. For patients with skeletal disease only, WHO criteria was used. For patients with measurable disease according to RECIST as well as bone metastasis, both RECIST & WHO were used.
  RECIST PD criteria required >=20% increase in certain target lesions OR progression of non-target lesions, or appearance of new lesions
  WHO PD criteria required increase in size of existing lesions or appearance of new lesions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Caelyx
Number analyzed (Participants) | 22
participants
  Patients followed by RECIST only (n=10) | 4
  Patients followed by WHO only (n=4) | 0
  Patients followed by RECIST & WHO (n=8) | 2

5. Secondary Outcome: Number of Patients Requiring Dose Reduction
Description: The protocol contains instructions to reduce the Caelyx dose according to specific schedules, in cases necessary due to reasons such as hematological toxicity, non-hematological toxicity, cardiotoxicity, or other toxic side-effects of treatment reducing quality of life etc.
Time Frame: Time of treatment until treatment discontinuation (study planned to continue until all participants ended treatment).
Measure: Number; unit: participants
Arm/Group | Caelyx
Number analyzed (Participants) | 25
participants
  Due to weight change | 6
  Due to toxicity/adverse event | 4

6. Secondary Outcome: Time to Response
Description: Response can be partial (>=30% decrease in the sum of Longest Diameter of target lesions, determined by two observations not less than 4 weeks apart; no unequivocal increase in the size of non-target lesions or the appearance of new lesions may occur) or complete (disappearance of all clinical evidence of tumor determined by 2 observations not less than 4 weeks apart), whichever status is recorded first.
Time Frame: Time of treatment until response, assessed every 12th week until end of treatment (study planned to continue until all participants ended treatment).
Population: Only 3 patients had measureable time to response
Measure: Median (Full Range); unit: Weeks
Arm/Group | Caelyx
Number analyzed (Participants) | 3
Weeks
  Patient 1 | 12.2 [12.2 to 12.2]
  Patient 2 | 11.4 [11.4 to 11.4]
  Patient 3 | 12.0 [12.0 to 12.0]

7. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time span from the first evaluation that shows response until the first evaluation that shows progression. Where patients did not show progress, duration of response was measured from the first evaluation that showed response until they discontinued the study.
  Response can be partial or complete (as previously defined), whichever status is recorded first.
Time Frame: as for outcome 2
Population: Three patients showed Partial Response according to RECIST criteria.
Measure: Median (Full Range); unit: weeks
Arm/Group | Caelyx
Number analyzed (Participants) | 3
weeks
  Patient 1 | 11.8 [11.8 to 11.8]
  Patient 2 | 48.6 [48.6 to 48.6]
  Patient 3 | 17.8 [17.8 to 17.8]

8. Secondary Outcome: Time to Progression
Description: Progression is defined as the first evaluation that shows progression (either by RECIST or WHO criteria):
  Progressive Disease according to RECIST response criteria: >=20% increase in the sum of the Longest Diameter of target lesions or unequivocal progression of non-target lesions. Appearance of new lesions will also constitute progressive disease.
  Progressive Disease according to WHO response criteria: Increase in size of existing lesions or appearance of new lesions.
Time Frame: Time of treatment until progression, assessed every 12th week until end of treatment (study planned to continue until all participants ended treatment).
Population: Of the 25 patients in the study 3 patients had non-measurable disease and could not be included in the progression analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Caelyx
Number analyzed (Participants) | 22
months | 5.69 [3.74 to 13.8]

9. Secondary Outcome: Duration of Overall Survival
Description: Patients were followed with regards to survival even after they left the trial (ie after End of Treatment visit). Deaths that occurred after patient participation ended were collected all the way through to the overall end of the trial which took place on Oct 31, 2009. These deaths were used to calculate overall survival.
Time Frame: Time of treatment until death, up to the time that all participants ended treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Caelyx
Number analyzed (Participants) | 25
months | 20.6 [6.58 to 25.6]

10. Secondary Outcome: Number of Days the Patients Were Hospitalized for Cancer-related Symptoms or Toxicity of Treatment
Description: The cumulative sum of hospitalization days during the study, per patient. Some patients had multiple hospitalizations.
Time Frame: Time of treatment until treatment discontinuation (study planned to continue until all participants ended treatment).
Population: Of the 25 total patients, 12 were hospitalized during the study.
Measure: Number; unit: days
Arm/Group | Caelyx
Number analyzed (Participants) | 12
days
  Patient 1 | 1
  Patient 2 | 1
  Patient 3 | 6
  Patient 4 | 4
  Patient 5 | 5
  Patient 6 | 71
  Patient 7 | 16
  Patient 8 | 1
  Patient 9 | 1
  Patient 10 | 3
  Patient 11 | 33
  Patient 12 | 20

ADVERSE EVENTS:
Time Frame: Time of treatment until treatment discontinuation (study planned to continue until all participants ended treatment).
Arm/Group | Caelyx
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx (N=25)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
PYREXIA (General disorders) | 2 (2)
CENTRAL LINE INFECTION (Infections and infestations) | 1 (1)
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 (1)
CYSTITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx (N=25)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (7)
DRY EYE (Eye disorders) | 2 (2)
LACRIMATION INCREASED (Eye disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (6)
CONSTIPATION (Gastrointestinal disorders) | 6 (7)
DIARRHOEA (Gastrointestinal disorders) | 6 (9)
FLATULENCE (Gastrointestinal disorders) | 2 (2)
GASTRITIS (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 16 (31)
STOMATITIS (Gastrointestinal disorders) | 6 (15)
VOMITING (Gastrointestinal disorders) | 7 (12)
CHEST PAIN (General disorders) | 3 (4)
FATIGUE (General disorders) | 17 (21)
OEDEMA PERIPHERAL (General disorders) | 4 (5)
PYREXIA (General disorders) | 6 (11)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 3 (3)
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 (4)
HAEMOGLOBIN DECREASED (Investigations) | 2 (2)
WEIGHT DECREASED (Investigations) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 9 (9)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (9)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)
DIZZINESS (Nervous system disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 (6)
BLISTER (Skin and subcutaneous tissue disorders) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (3)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 13 (18)
RASH (Skin and subcutaneous tissue disorders) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish data from the study, a copy must be provided to the sponsor for review at least 60 days before submission for publication. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days. If issues arise regarding scientific integrity or regulatory compliance, the sponsor will review these issues with the investigator. The sponsor will not change scientific content or suppress information.